CLINICAL TRIAL: NCT02259582
Title: A 2-Arm Phase 2 Double-Blind Randomized Study of Carboplatin, Pemetrexed Plus Placebo Versus Carboplatin, Pemetrexed Plus Truncated Demcizumab as First-Line Treatment in Subjects With Stage IV Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Carboplatin, Pemetrexed Plus Placebo vs Carboplatin, Pemetrexed Plus 1 or 2 Truncated Courses of Demcizumab in Subjects With Non-Squamous Non-Small Cell Lung Cancer
Acronym: DENALI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M18-007
Record Dates: First submitted 2014-09-17; First posted 2014-10-08 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Nonsquamous Nonsmall Cell Neoplasm of Lung
Keywords: Phase 2; histologically; confirmed; malignancy; metastatic; pemetrexed; carboplatin; carcinoma; non small cell lung; lung neoplasms; lung diseases
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Carcinoma; Lung Neoplasms; Lung Diseases | interventions — Pemetrexed; Carboplatin; demcizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 Pem, carbo, placebo x 4 cycles (Placebo Comparator): Pemetrexed (500 mg/m2),carboplatin (area under the concentration-time curve of 6 mg/mL x min) once every 21 days X 4 cycles, pemetrexed maintenance and placebo starting at Day 84
  Interventions: Drug: Pemetrexed; Drug: Carboplatin
- Arm 2 Pem, carbo x 4 cycles, one course of dem (Active Comparator): Pemetrexed (500 mg/m2), carboplatin (area under the concentration-time curve of 6 mg/mL x min) x 4 cycles, one course of demcizumab 5mg/kg, maintenance pemetrexed + placebo starting on Day 84
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: demcizumab
- Arm 3 pem, carbo, dem x 4 cycles, dem retreatment (Active Comparator): Pemetrexed (500 mg/m2), carboplatin (area under the concentration-time curve of 6 mg/mL x min) x 4 cycles, maintenance pemetrexed starting on Day 84. 2 courses of demcizumab 5 mg/kg
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: demcizumab

INTERVENTIONS:
Drug: Pemetrexed
Drug: Carboplatin
Drug: demcizumab
  Arms: Arm 2 Pem, carbo x 4 cycles, one course of dem; Arm 3 pem, carbo, dem x 4 cycles, dem retreatment

SUMMARY:
A randomized, double-blind, 3-arm (1:1:1) study in subjects with first-line Stage IV non-squamous NSCLC. The purpose is to test the efficacy and safety of demcizumab, when given in combination with carboplatin and pemetrexed compared to placebo. The administration of carboplatin and pemetrexed is a standard treatment for patients with non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
Patients will be enrolled at centers in North America, Western Europe, Australia and New Zealand. Up to 28 days (4 weeks) prior to treatment.

If enrolled in the study, you will receive intravenous (in the vein) infusions of demcizumab (or placebo), carboplatin, and pemetrexed administered on the same day, every 21 days for 4 cycles, or until it has been shown that your cancer has gotten worse. If your physician decides to delay treatment with one of the agents due to side effects, the other agents may still be administered as scheduled. After 4 cycles, if you have stable or improved disease, you will continue to receive pemetrexed once every 21 days as maintenance therapy. After 8 cycles, if you have stable or improved disease, you may receive demcizumab (or placebo), every 21 days for 4 more cycles.

You will undergo assessments every 6 weeks to determine the status of your disease.

ELIGIBILITY:
Main Inclusion Criteria:

1. Signed Informed Consent Form
2. Histologically or cytologically confirmed Stage IV non-squamous NSCLC
3. Availability of FFPE (formalin-fixed paraffin-embedded) tumor tissue, either fresh core-needle-biopsied or archived
4. Age > or = to 21 years
5. ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1
6. Disease that is measurable per RECIST v1.1
7. Adequate organ and marrow function
8. For women of childbearing potential, agreement to use two effective forms of contraception

Main Exclusion Criteria:

1. Histologically or cytologically documented, advanced, mixed non-small cell and small cell tumors or mixed adenosquamous carcinomas
2. NSCLC with known EGFR (epidermal growth factor receptor ) mutation or anaplastic lymphoma kinase (ALK) gene translocation (such as EML4 [echinoderm microtubule-associated protein-like 4]-ALK [anaplastic lymphoma kinase])
3. Prior or ongoing therapy (including chemotherapy, antibody therapy, tyrosine kinase inhibitors, radiotherapy, immunotherapy, hormonal therapy, or investigational therapy) for the treatment of Stage IV non-squamous NSCLC
4. Evidence of tumor invading major blood vessels, cavitation of one or more pulmonary tumor mass(es) or tracheo-esophageal fistula
5. Brain metastases, leptomeningeal disease, uncontrolled seizure disorder, or active neurologic disease
6. Malignancies other than non-squamous NSCLC successfully treated within 3 years prior to randomization (with the exception of certain early-stage cancers)
7. History of a significant allergic reaction attributed to humanized or human monoclonal antibody therapy
8. Significant intercurrent illness defined as an illness that may result in the subject's death prior to their death from non-squamous NSCLC and/or significantly limit their ability to comply with the requirements of this study
9. Recent hemoptysis >2.5 mL or serious bleeding from another site, known bleeding disorder or coagulopathy or therapeutic anti-coagulation
10. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization, or anticipation of need for major surgical procedure during the course of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (18):
  - Desert Hematology Oncology Medical Group, Inc., Rancho Mirage, California
  - University of California, San Francisco, San Francisco, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Ocala Oncology Center, Ocala, Florida
  - Edward H. Kaplan MD & Associates, Skokie, Illinois
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Broome Oncology, LLC, Binghamton, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Gaston Hematology & Oncology, Gastonia, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Texas Oncology-Sherman, Sherman, Texas
  - Compass Oncology, Vancouver, Washington
- Australia (8):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - The Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - North Coast Cancer Institute Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Royall Brisbane & Women's Hospital, Herston, Queensland
  - Icon Cancer Foundation, Milton, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Monash Health, Monash Cancer Centre-Moorabbin, Bentleigh East, Victoria
  - St. John of God Subiaco Hospital, Subiaco, Western Australia
- Belgium (4):
  - Ziekenhuisnetwerk Antwerpen- Koningin Paola Kinderzickenhuis, Antwerp
  - Grand Hopital de Charleroi- Site Notre-Dame, Charleroi
  - Centre Hospitalier Jolimont-Lobbes, La Louvière
  - CHR de Ia Citadelle, Liège
- Italy (4):
  - Azienda Ospedaliera Istituti Ospitalieri, Cremona, Lombardy
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Smilow Cancer Hospital at Yale-New Haven, Aviano, Pordenone
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
- Spain (11):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Nuestra Senora de Sonsoles, Ávila
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institute Catalan de Oncologia (ICO L'Hospitalet), Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Madrid Universitario Sanchinarro, Madrid
  - Hospital Universitario Virgen del Rocio, Seville

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Placebo Arm (Arm 1): Placebo plus pemetrexed and carboplatin (4 cycles), pemetrexed (4 cycles), placebo plus pemetrexed (4 cycles)
- Demcizumab/Placebo Arm (Arm 2): Demcizumab plus pemetrexed and carboplatin (4 cycles), pemetrexed (4 cycles), placebo plus pemetrexed (4 cycles)
- Demcizumab/Demcizumab Arm (Arm 3): Demcizumab plus pemetrexed and carboplatin (4 cycles), pemetrexed (4 cycles), demcizumab plus pemetrexed (4 cycles)
Period: Overall Study
Arm/Group | Placebo/Placebo Arm (Arm 1) | Demcizumab/Placebo Arm (Arm 2) | Demcizumab/Demcizumab Arm (Arm 3)
Started | 25 | 28 | 29
Completed | 9 | 11 | 8
Not Completed | 16 | 17 | 21
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Disease progression | 14 | 15 | 17
Not completed — Lack of Subject Adherence to Protocol | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Placebo Arm (Arm 1) | Demcizumab/Placebo Arm (Arm 2) | Demcizumab/Demcizumab Arm (Arm 3) | Total
Number analyzed (Participants) | 25 | 28 | 29 | 82
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 77] | 66 [31 to 76] | 61 [39 to 76] | 62 [31 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 12 | 42
  Male | 10 | 13 | 17 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 23 | 26 | 28 | 77
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 1 | 1 | 2
  United States | 5 | 8 | 7 | 20
  Italy | 2 | 2 | 3 | 7
  Australia | 14 | 10 | 10 | 34
  Spain | 4 | 7 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Investigator-assessed (RECIST) v1.1 Response Rate in the Treatment Arms.
Description: Investigator-assessed Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 response rate (unconfirmed) in placebo/placebo arm to demcizumab/placebo arm and demcizumab/demcizumab arm combined in subjects with first-line stage IV non-small cell lung cancer (NSCLC). Response rate was based on Investigator-assessed best-overall-response (BOR) and was defined as the best unconfirmed response determined by RECIST version 1.1 recorded from the start of the treatment until disease progression in the following order of importance: CR, PR , SD, progressive disease (PD), not evaluable, or missing.
Time Frame: Response assessment data was collected until the subject started alternative anti-cancer treatment or developed progressive disease, whichever occurred first, assessed up to approximately 26 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Placebo Arm (Arm 1) | Demcizumab/Placebo Arm (Arm 2) | Demcizumab/Demcizumab Arm (Arm 3)
Number analyzed (Participants) | 25 | 28 | 29
Participants
  Complete response (CR) | 0 | 0 | 0
  Partial response (PR) | 13 | 10 | 6
  Stable disease (SD) | 10 | 14 | 15
  Progressive disease (PD) | 2 | 4 | 5
  Not evaluable (NE) | 0 | 0 | 0
  Missing | 0 | 0 | 3
Statistical Analysis 1: Comparison: Placebo/Placebo Arm (Arm 1) vs Demcizumab/Placebo Arm (Arm 2) vs Demcizumab/Demcizumab Arm (Arm 3); The Kaplan-Meier method was used to estimate both the survival curves and the median survival time. The 95% confidence interval (CI) for the median survival time was calculated. A p-value for treatment effect was generated using a stratified Cox proportional hazards model; Test type: Superiority — Based on RECIST v1.1. Response outcomes from an assessment done anytime less than Day 35 were considered as not evaluable unless the response assessment was progress disease; p = 0.0401, Log Rank; Hazard Ratio (HR) = 0.04, 95% CI 2-sided [.013 to .095]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at every weekly study visit from randomization until 30 days after the termination visit for up to approximately 26 months.
Description: All reported adverse events were mapped to standard MedDRA coding terms, grouped by system organ class and preferred term and tabulated by treatment arm.
Arm/Group | Placebo/Placebo Arm (Arm 1) | Demcizumab/Placebo Arm (Arm 2) | Demcizumab/Demcizumab Arm (Arm 3)
All-Cause Mortality (participants affected / at risk) | 1/25 | 2/28 | 2/29
Serious Adverse Events (participants affected / at risk) | 6/25 | 11/28 | 15/29
Other Adverse Events (participants affected / at risk) | 25/25 | 28/28 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Placebo Arm (Arm 1) (N=25) | Demcizumab/Placebo Arm (Arm 2) (N=28) | Demcizumab/Demcizumab Arm (Arm 3) (N=29)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 2 (2) — administration site conditions
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Placebo Arm (Arm 1) (N=25) | Demcizumab/Placebo Arm (Arm 2) (N=28) | Demcizumab/Demcizumab Arm (Arm 3) (N=29)
Hypertension (Vascular disorders) | 4 (4) | 14 (14) | 12 (12)
Hypotension (Vascular disorders) | 4 (4) | 2 (2) | 3 (3)
Fatigue (General disorders) | 15 (15) | 16 (16) | 12 (12)
Asthenia (General disorders) | 8 (8) | 10 (28) | 9 (29)
Pyrexia (General disorders) | 4 (4) | 6 (6) | 9 (9)
Oedema peripheral (General disorders) | 5 (5) | 4 (4) | 1 (1)
Malaise (General disorders) | 3 (3) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 5 (5) | 7 (7)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 8 (8) | 6 (6)
Alanine aminotransferase increased (Investigations) | 6 (6) | 4 (4) | 3 (3)
Platelet count decreased (Investigations) | 4 (4) | 4 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 3 (3) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (3) | 3 (3) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2) | 3 (3) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 11 (11) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 6 (6) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 7 (7) | 11 (11) | 7 (7)
Dizziness (Nervous system disorders) | 8 (8) | 9 (9) | 2 (2)
Dysgeusia (Nervous system disorders) | 8 | 3 | 2
Lacrimation increased (Eye disorders) | 3 (3) | 5 (5) | 3 (3)
Dry eye (Eye disorders) | 3 (3) | 3 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 18 (18) | 18 (18) | 14 (14)
Constipation (Gastrointestinal disorders) | 15 (15) | 11 (11) | 11 (11)
Vomiting (Gastrointestinal disorders) | 9 (9) | 8 (8) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 6 (6) | 13 (13)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 4 (4) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 4 (4) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 11 (11) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT02259582/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT02259582/Prot_ICF_001.pdf